CLINICAL TRIAL: NCT02686424
Title: Tumor Markers Study in Gastric Cancer for Cancer Immunotherapy
Brief Title: Tumor Markers Study in Gastric Cancer for Cancer Immunotherapy (ONCO-RD 010 CRT)
Acronym: ONCO-RD010CRT
Status: Suspended | Type: Observational
Why Stopped: paperwork delay
Sponsor: Seoul National University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Woo Ho Kim, Professor, Seoul National University Hospital
Other Study IDs: ONCO-RD 010 CRT (114824)
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Stomach Neoplasms
Keywords: MAGE-A3 protein; NY-ESO-1 protein; WT1 Proteins; PRAME protein
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Gastric cancer is one of the leading causes of cancer-related deaths worldwide. Despite advances in therapeutic intervention, the mortality from this disease remains high. As a result, most patients are now offered varying combinations of surgery, chemotherapy, and radiation therapy in order to derive benefits from a multidisciplinary approach. Unfortunately, therapies are often toxic or debilitating and therapeutic responses can vary. Thus new therapeutic strategy is required for the treatment of gastric cancer.

In the early 1980s, the discovery of cytolytic T cells (cytolytic T lymphocytes, CTLs) directed against an antigen presented on tumor cells was published. They can kill many invasive cells by recognizing the tumor specific antigens on the major histocompatibility complex (MHC) molecules. It is now generally agreed that although tumors express tumor antigens, they usually lack immunogenicity because of their inability to activate the immune response. The current view is that tumor cells are antigenic, but not immunogenic. If we can artificially activate the immune system against the tumor, it may be possible to eradicate the tumor. This approach is the basis of cancer immunotherapy.

Many tumor antigens have been defined in terms of multiple solid tumors: MART-1/Melan-A, gp100, carcinoembryonic antigen (CEA), HER-2, mucins (i.e., MUC-1), prostate-specific antigen (PSA), and prostatic acid phosphatase (PAP) are just a short list. Some immune-based therapies targeting these tumor antigens are in phase III trials assessing whether immunizing against these antigens affects overall survival. In gastric cancer, some tumor antigens such as MAGE-A3, NY-ESO-1, and WT-1 have been reported to be expressed in substantial proportion of cases. They have the potential to be the targeting molecules for immunotherapy in the future. In this study, we aim to explore the expression levels of the four tumor markers (MAGE-A3, NY-ESO-1, WT-1 and PRAME) in gastric cancers of Korean patients and to examine the correlations of the expression levels of the four markers to clinic-patholoical factors.

ELIGIBILITY:
Inclusion Criteria:

* gastric carcinoma
* received gastrectomy

Exclusion Criteria:

* neoadjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastric carcinoma patients who received ghastrectomy
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
overall survival | five years

IPD SHARING:
Plan to Share IPD: No